CLINICAL TRIAL: NCT00831077
Title: Pharmacokinetic Properties of ORM-14540 and ORM-12741 After Administration of a Microdose of 14C-labelled Drug; An Open, Non-randomised, Single Dose, Single Centre Study in Healthy Male Subjects
Brief Title: Early Phase I Microdosing Study of ORM-14540 and ORM-12741
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Mononen/Clinical Study Manager, Development
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3101001
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — ORM-12741

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 14C-ORM-14540 (Active Comparator)
  Interventions: Drug: ORM-14540
- 14C-ORM-12741 (Active Comparator)
  Interventions: Drug: ORM-12741

INTERVENTIONS:
Drug: ORM-14540 — i.v.
  Arms: 14C-ORM-14540
Drug: ORM-12741 — i.v.
  Arms: 14C-ORM-12741

SUMMARY:
The purpose of this study is to determine pharmacokinetic parameters of ORM-12741 and ORM-14540 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Good general health ascertained by detailed medical history and physical examinations.
* Males between 18 and 45 years (inclusive).
* Body Mass Index (BMI) between 18-30 kg/m2 (inclusive, BMI = weight/height2).
* Weight 55-100 kg (inclusive).

Exclusion Criteria:

* A predictable poor compliance or inability to communicate well with the investigator or study centre personnel.
* Veins unsuitable for repeated venipuncture
* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric diseases as judged by the investigator.
* Any condition requiring regular concomitant medication including herbal products or likely to need any concomitant treatment during the study.
* Susceptibility to severe allergic reactions.
* Intake of any medication that could affect the outcome of the study, within 2 weeks prior to the first study treatment or less than 5 times a half-life of the medication. Possible enzyme inducing drugs will be discussed case-by-case with the sponsor.
* Regular consumption of more than 21 units of alcohol per week (1 unit = 4 cl spirits, about 13 g of alcohol).
* Current use of nicotine-containing products more than 5 cigarettes or equivalent/day.
* Inability to refrain from using nicotine-containing products during the stay at the study centre.
* Inability to refrain from consuming caffeine-containing beverages during the stay in the study centre, e.g. propensity in getting headache when refraining from caffeine-containing beverages.
* Blood donation or loss of significant amount of blood within 2 months prior to the screening visit.
* Abnormal 12-lead electrocardiogram (ECG) finding of clinical relevance in supine position after resting for 10 minutes at the screening visit, for example:- QTc (calculated through the Bazett's formula) > 450msec,- PR < 120 msec or > 210 msec,- QRS < 70 msec or > 120 msec.
* Heart rate (HR) < 45 beats/minute or > 100 beats/minute in supine position after resting for 10 minutes at the screening visit.
* At the screening visit, systolic blood pressure (BP) < 90 mmHg or > 140 mmHg in supine position after resting for 10 minutes, diastolic BP < 50 mmHg or > 90 mmHg in supine position after resting for 10 minutes.
* Any abnormal value of laboratory, vital signs, or physical examination, which may in the opinion of the investigator interfere with the interpretation of the test results or cause a health risk for the subject if he takes part into the study.
* History of drug abuse or positive result in drug abuse test.
* Positive serology to human immunodeficiency virus antigen/antibodies (HIVAgAb), hepatitis C virus antibodies (HCVAb) or hepatitis B surface antigen (HBsAg).
* Any other condition that in the opinion of the investigator would interfere with the evaluation of the results or constitute a health risk for the subject.
* Participation in a clinical drug study within 3 months prior to the screening visit in this study, or earlier participation in a clinical study with ORM-12741.
* Exposure to 14C-labelled drugs or diagnostics within 12 months prior to the screening visit.
* Men who are not practising clinically accepted method of contraception during the study and next 3 months after the study treatment administration.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables including: Area under the concentration-time curve (AUC), Maximum observed concentration (Cmax) at the end of infusion, Terminal elimination half-life (t½z), Total clearance (CL) | 72 hours

SECONDARY OUTCOMES:
Safety variables including blood pressure (BP), heart rate (HR), electrocardiograms (ECGs), physical examination, laboratory safety variables (haematology, chemistry, serology and urinalysis) and adverse events (AEs). | Before and after study

CONTACTS AND LOCATIONS:
Overall Officials: Juha Peltonen, MD, Principal Investigator — CRST; Virpi Mononen, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- CRST, Turku, Finland